CLINICAL TRIAL: NCT02026791
Title: The Comparison of the Clinical Efficacy Between I-gel and LMA-Supreme, the Two Most Recently Developed Supraglottic Airway Devices, in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4-2013-0723
Record Dates: First submitted 2013-12-18; First posted 2014-01-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: The Elderly Patients Aged Between 65 and 85
Keywords: Supraglottic airway device; I-gel; SupremeLMA; Elderly patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The clinical efficacy of the I-gel (Experimental): The clinical efficacy of the I-gel
  Interventions: Device: I-gel
- The clinical efficacy Supreme-LMA (Active Comparator): The clinical efficacy Supreme-LMA
  Interventions: Device: Supreme-LMA

INTERVENTIONS:
Device: I-gel — * The patient was monitored at 1-5 minute intervals.
  * While supplying oxygen through a mask, propofol 1.0mg/kg and remifentanil 0.5ug/kg were intravenously injected to induce anesthesia. When consciousness was not lost, propofol 0.5mg/kg was additionally injected. After consciousness was lost and spontaneous respiration disappeared, rocuronium 0.3 mg/kg was intravenously injected while performing manual ventilation.
  * After injecting an anesthetic and muscle relaxant, the injection concentration of fresh gas including 6 L/min oxygen and desflurane was regulated to maintain BIS between 40 and 60. A train of four (TOF) was performed with a nerve stimulator for muscle relaxation monitoring to verify that a muscular contraction did not take place (TOF=0).
  * Then, with the assistance of another anesthesiologist, I-gel prepared in advance was inserted.
  Arms: The clinical efficacy of the I-gel
Device: Supreme-LMA — * The patient was monitored at 1-5 minute intervals.
  * While supplying oxygen through a mask, propofol 1.0mg/kg and remifentanil 0.5ug/kg were intravenously injected to induce anesthesia. When consciousness was not lost, propofol 0.5mg/kg was additionally injected. After consciousness was lost and spontaneous respiration disappeared, rocuronium 0.3 mg/kg was intravenously injected while performing manual ventilation.
  * After injecting an anesthetic and muscle relaxant, the injection concentration of fresh gas including 6 L/min oxygen and desflurane was regulated to maintain BIS between 40 and 60. A train of four (TOF) was performed with a nerve stimulator for muscle relaxation monitoring to verify that a muscular contraction did not take place (TOF=0).
  * Then, with the assistance of another anesthesiologist, Supreme LMA prepared in advance was inserted.
  Arms: The clinical efficacy Supreme-LMA

SUMMARY:
Since the laryngeal mask airway (LMA) was designed and introduced into a clinical setting, a supraglottic airway device is widely used because it has advantages such as manipulation of the device when inserting it is easier than that of an endotracheal tube and it causes less postoperative sore throats. Insertion of an LMA can be performed relatively easily and safety at an appropriate depth of anesthesia when compared with the insertion of an endotracheal tube because an LMA is inserted without using a laryngoscope and without causing stimulus to the vocal cords and the trachea. Hence, an LMA may be useful in cases of coronary artery disease and a carotid endarectomy where stabilization of the cardiopulmonary function is important. In addition, an LMA is hemodynamically stable not only in the induction of anesthesia but also in the arousal of anesthesia and thus less dangerous to a cardiovascular disease patient. LMA may be useful also to patients having chronic obstructive lung disease because the patients have an excessively sensitive airway and ventilation is difficult to perform in them. Therefore, in elderly patients having a prevalence for cardiovascular disease or chronic obstructive lung disease, use of an LMA, which stimulates the airway less, may provide hemodynamical stability and reduce relevant complications or side effects. LMA Supreme which is newly designed in such ways has been proven to be superior to the conventional LMA Classic in terms of easy insertion and oropharyngeal sealing. A study which compared LMA Classic and LMA Supreme with adult subjects showed that LMA Supreme had a superior insertion success rate and better oropharyngeal leak pressure (OLP) than those of LMA Classic. Another newly developed supraglottic airway device is I-gel. In I-gel, which is a disposable, latex-free LMA, a soft, gel-type cuff made of a thermoplastic elastomer replaces the inflatable cuff of other LMAs. Thus, I-gel has an advantage that, once it is installed, it requires no additional clinical manipulation such as cuff inflation or cuff pressure monitoring. A comparison of I-gel with LMA Classic and other disposable supraglottic airway devices produced by various manufactures in adult subjects showed that the clinical properties were similar with respect to easy insertion, time required for installation, laryngopharynx leak pressure, and degree of glottis exposure observed with a fiberoptic bronchoscope. Thus, I-gel is expected to be a supraglottic airway device which may replace the conventional LMA Classic. The elderly are known to have an upper airway anatomically different from that of younger adults depending on age. A study conducted with CT showed that normal elderly people had a wider upper airway than that of younger males or middle-aged males and that elderly with accompanying sleep apnea had a wider upper airway than that of younger males in all regions including the nasopharynx, oropharynx, and hypopharynx. Therefore, because the upper airway of the elderly is wider and longer, a different supraglottic airway device guide may be necessary. Our previous studies showed that the single time success rate was significantly lower, the insertion was more difficult, and the insertion took a longer time when the LMA classic was used in elderly patients than in younger adult patients. However, there is no available guide for the use of a supraglottic airway device or for a supraglottic airway device more appropriate for elderly patients. Moreover, no study has been ever conducted with regard to such a guide.

Therefore, in this study, the clinical usefulness of I-gel and LMA Supreme, which are the newest supraglottic airway devices, was verified in elderly patients. It was also verified which of the two devices is better to use as a supraglottic airway device.

ELIGIBILITY:
Inclusion Criteria:

* The elderly patients aged between 65 and 85
* The patient having a plan for a regular operation under general anesthesia in which the expected operation duration is within two hours and the airway may be managed intraoperatively with a supraglottic airway device.

Exclusion Criteria:

* The patients having an anatomical structure which may cause difficulty in mask respiration
* The patients having an upper airway infection or an airway-related disease such as asthma and pneumonia.
* The patients having a risk of aspiration such as gastroesophageal reflux.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The success insertion rate of supraglottic airway devices of the first trial was the primary end point. | Average 10 seconds after induction and during average 10 mins
  The success insertion rate of supraglottic airway devices of the first trial was the primary end point. In success insertion of supraglottic airway devices is confirmed by following cases of manual ventilation.
  1. Appropriateness of the chest wall movement
  2. A square wave in the capnograph
  3. The time taken until the successful installation of an LMA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Kim MH, Lee JH, Choi YS, Park S, Shin S. Comparison of the laryngeal mask airway supreme and the i-gel in paralysed elderly patients: A randomised controlled trial. Eur J Anaesthesiol. 2018 Aug;35(8):598-604. doi: 10.1097/EJA.0000000000000700. PMID 28857785